CLINICAL TRIAL: NCT03733691
Title: A Phase 2, Open Label, Randomized Trial Evaluating Ixazomib Compared to Ixazomib-Lenalidomide Combination Maintenance Therapy for Frontline Multiple Myeloma Patients
Brief Title: Ph 2 Maintenance Trial: Ixazomib vs Ixazomib-Lenalidomide for MM Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Oncotherapeutics (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X16108
Record Dates: First submitted 2018-11-02; First posted 2018-11-07 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Newly Diagnosed Multiple Myeloma
Keywords: Multiple Myeloma; Front-line; Maintenance therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Lenalidomide

STUDY DESIGN:
Intervention Model Description: A randomized, open label, Phase 2 study involving two arms evaluating the efficacy and safety of ixazomib monotherapy (with steroids if applicable) and the combination of ixazomib and lenalidomide (with steroids if applicable) as maintenance therapy for patients with MM who have achieved at least PR after receiving a bortezomib and lenalidomide (with steroids if applicable)-containing combination frontline therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ixazomib Only (Experimental): The prescribed dose administration of ixazomib in this study is 3mg orally on Days 1, 8, and 15 of a 28-day cycle.
  Interventions: Drug: Ixazomib
- Ixazomib + Lenalidomide (Experimental): The prescribed dose administration of ixazomib in this study is 3mg orally on Days 1, 8, and 15 of a 28-day cycle.
  The prescribed dose administration of lenalidomide in this study is the same as the dose of the patient's front-line treatment taken in the last treatment cycle unless otherwise clinically indicated per investigator's discretion, taken orally on days 1-28 of a 28-day cycle. If patient was receiving lenalidomide at a higher dose than 10 mg, then the dose of lenalidomide on this study will be adjusted to 10 mg daily on days 1-28 of a 28-day cycle
  Interventions: Drug: Ixazomib; Drug: Lenalidomide

INTERVENTIONS:
Drug: Ixazomib — 3 mg oral capsule, Days 1, 8 and 15 of 28-day cycles
  Other Names: Ninlaro
Drug: Lenalidomide — Same dose as in the front-line treatment in the last treatment cycle, taken orally, on days 1-28 of a 28-day cycle.
  Other Names: Revlimid
  Arms: Ixazomib + Lenalidomide

SUMMARY:
This is a randomized, Phase 2 study involving two arms evaluating the efficacy and safety of ixazomib alone and the combination of both ixazomib and lenalidomide as maintenance therapy for patients with multiple myeloma who have achieved at least partial response (PR) or better after receiving a bortezomib- and lenalidomide-containing combination front-line therapy.

DETAILED DESCRIPTION:
Patients who have achieved PR or better on a bortezomib- and lenalidomide-containing combination therapy will be randomized to receive maintenance therapy with 28-day cycles of either ixazomib alone or the combination of ixazomib and lenalidomide. If steroids were part of the patient's qualifying regimen, steroids will be administered using the same drug(s), schedule(s) and dose(s) as those of the last treatment cycle of the bortezomib-, lenalidomide- and steroid-containing regimen. Ixazomib will be administered per orem (PO) at 3 mg on days 1, 8 and 15 of 28-day cycles. Lenalidomide will be taken PO, once daily at the same dose as the last treatment on days 1 through 28 of the 28-day cycles. Patients will start the randomized maintenance therapy after receiving a minimum of 6 cycles of a bortezomib- and lenalidomide-containing combination treatment but may have received up to 8 cycles if they continued to show improvement in their response after the first 6 cycles. During cycle 1, patients will have clinical laboratory tests weekly (days 1, 8, 15 and 22) and MM disease assessments on day 22 to monitor for efficacy and potential toxicity. Beginning with cycle 2, patients will have clinical laboratory tests performed twice a month and MM disease assessments once a month. Patients will be treated until documentation of PD or if subject meets any of the treatment discontinuation criteria.

ELIGIBILITY:
Inclusion Criteria:

-

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

1. Male or female patients 18 years or older.
2. Patients must be receiving a frontline bortezomib- and lenalidomide-containing regimen for treatment of disease
3. Patients must meet the following clinical laboratory criteria:

   * Absolute neutrophil count (ANC) grater or equal 1,000/mm3 and platelet count greater or equal 75,000/mm3. Platelet transfusions to help patients meet eligibility criteria are not allowed within 7 days prior to screening platelets or at investigator's discretion.
   * Hemoglobin ≥ 8.0 g/dL. Use of erythropoietic stimulating factors and red blood cell (RBC) transfusions per institutional guidelines is allowed; however, most recent RBC transfusion must have been at least 7 days prior to obtaining screening hemoglobin or at investigator's discretion.
   * Total bilirubin less or equal 1.5 times the upper limit of the normal range (ULN).
   * Calculated or measured creatinine clearance greater or equal 30 mL/min. Calculation is based on a standard Cockcroft and Gault formula (Section 14.2).
   * AST (SGOT) and ALT (SGPT) less or equal 3 x ULN or less or equal 5 x ULN if hepatic metastases are present.
   * LVEF ≥ 40%. 2-D transthoracic echocardiogram (ECHO) is the preferred method of evaluation. Mitigated Acquisition Scan (MUGA) is acceptable if ECHO is not available.
4. Patients must be transplant ineligible as determined by the treating physician.
5. Patients must have a life-expectancy of more than 6 months.
6. Patients must have a confirmed diagnosis of MM.
7. Patients receiving front-line therapy must have achieved at least PR and have completed at least 6 cycles of treatment.
8. The disease must have reached a plateau phase at the end of front-line treatment as demonstrated bythe same response (using IMWG criteria) in three consecutive tests with at least three weeks between each test.
9. Patients must have received frontline treatment within 8 weeks of enrollment.
10. Patient can adhere to the study visit schedule and other protocol requirements.
11. Patient Eastern Cooperative Oncology Group (ECOG) performance status is ≤ 2.
12. Patients must voluntarily give written consent before any study related procedure not part of standard medical care is performed, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
13. Female patients must be postmenopausal for at least 1 year before screening visit OR surgically sterile. If patient is female of childbeating potential (FCBP), patient must agree to practice two effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug. FCBP must also adhere to the guidelines of any treatment-specific pregnancy prevention program AND agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
14. Male patients, even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

    * To practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug
    * To practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

* Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

  1. Patient is currently progressing on a bortezomib- and lenalidomide-containing regimen.
  2. Patients who have received more than 1 line of therapy (thus non-frontline treated patients).
  3. Patients who were exposed to ixazomib during frontline therapy.
  4. Patient has ¬> Grade 3 peripheral neuropathy or Grade 2 with pain during the screening period.
  5. Patient has known gastrointestinal disease or gastrointestinal procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing.
  6. Female patients who are lactating or have a positive serum pregnancy test during the screening period.
  7. Major surgery within 14 days before enrollment or at investigator's discretion.
  8. Patients undergoing stem cell therapy (SCT) or those who are planned for SCT.
  9. Radiotherapy within 14 days before enrollment or investigator's discretion. If the involved field is small, 7 days or investigator's discretion will be considered a sufficient interval between treatment and administration of the study drugs. Receipt of localized radiation therapy does not preclude enrollment.
  10. Infection requiring systemic antibiotic therapy or other serious infection such as known active hepatitis B or C virus infection, known human immunodeficiency virus (HIV) positive within 14 days before of study enrollment or at investigator's discretion.
  11. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, NYHA Class III or IV heart failure, unstable angina, clinically significant pericardial disease or myocardial infarction within the past 6 months, unless subject has a pacemaker. Prior to study entry, any ECG abnormality at Screening must be documented by the investigator as not medically relevant.
  12. Frontline therapy within 14 days or at investigator's discretion of the first dose of study drugs.
  13. Systemic treatment, within 14 days before or at investigator's discretion of the first dose of study drugs, with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort or Ginkgo biloba.
  14. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
  15. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
  16. Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease.

      • Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
  17. Participation in other clinical trials throughout the duration of this trial.
  18. Patient has been diagnosed with:

      1. Plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M protein) and skin changes (POEMS) syndrome3.
      2. Primary amyloidosis
      3. Plasma cell leukemia.
      4. Severe hypercalcemia, i.e., serum calcium ≥ 12 mg/dL (3.0 mmol/L) corrected for albumin.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
PFS | Through study completion, approximately 5 years
  Progression Free Survival
Adverse events (AEs) | throughout the study completion, approximately 5 years
  Monitoring safety and tolerability via monitoring adverse events graded by CTCAE v5

SECONDARY OUTCOMES:
OS | from time of initiation of maintenance therapy to death from any cause or last follow-up visit, up to 60 months
  Overall survival
Deepening of the response | throughout the study, up to 60 months
  define as the percentage of patients who improved their response during maintenance therapy.

CONTACTS AND LOCATIONS:
Overall Officials: James R. Berenson M Inc., MD, Principal Investigator — Oncotherapeutics
Locations (1):
- James R Berenson, MD, Inc., West Hollywood, California, United States

IPD SHARING:
Plan to Share IPD: No